CLINICAL TRIAL: NCT04708041
Title: A Phase 3 International, Multicenter, Open-label Study to Evaluate the Safety and Immunogenicity of 9vHPV Vaccine Administered as 2-dose Regimen With Extended Dosing Intervals in 9- to 14-Year Old Boys and Girls Compared With a Standard 3-dose Regimen in 16- to 26-Year Old Women
Brief Title: Safety and Immunogenicity of Extended 2-dose Regimens of 9-valent Human Papillomavirus (9vHPV) Vaccine (V503-069)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-069; V503-069 (Other: MSD); 2022-500253-37 (Registry Identifier: EU CT); U1111-1274-2496 (Registry Identifier: UTN); 2020-003736-24 (EudraCT Number)
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 0: 1 Dose of 9vHPV Vaccine (previous 1-dose recipients) (Experimental): 10 to 15 year old girls and boys (who previously received 1 dose of 9vHPV vaccine) receive a second dose of 9vHPV vaccine at Day 1.
  Interventions: Biological: 9vHPV vaccine
- Cohort 1: 2 Doses of 9vHPV Vaccine Given 12 Months Apart (Experimental): 9 to 14 year old girls and boys receive a 2-dose regimen of 9vHPV vaccine at Day 1 and Month 12.
  Interventions: Biological: 9vHPV vaccine
- Cohort 2: 2 Doses of 9vHPV Vaccine Given 24 Months Apart (Experimental): 9 to 13 year old girls and boys receive a 2-dose regimen of 9vHPV vaccine at Day 1 and Months 24.
  Interventions: Biological: 9vHPV vaccine
- Cohort 3: 2 Doses of 9vHPV Vaccine Given 36 Months Apart (Experimental): 9 to 12 year old girls and boys receive a 2-dose regimen of 9vHPV vaccine at Day 1 and Month 36.
  Interventions: Biological: 9vHPV vaccine
- Cohort 4: 2 Doses of 9vHPV Vaccine Given 60 Months Apart (Experimental): 9 to 10 year old girls and boys receive a 2-dose regimen of 9vHPV vaccine at Day 1 and Month 60.
  Interventions: Biological: 9vHPV vaccine
- Cohort 5: 3 Doses of 9vHPV Vaccine Given Over a 6-Month Period (Active Comparator): 16 to 26 year old young women receive 3 dose regimen of 9vHPV vaccine at Day 1, Month 2 and Month 6.
  Interventions: Biological: 9vHPV vaccine

INTERVENTIONS:
Biological: 9vHPV vaccine — 9-valent human papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) administered as a 0.5-mL intramuscular injection

SUMMARY:
This is a 96-month safety and immunogenicity study conducted in boys and girls 9 to 14 years of age and in young women 16 to 26 years of age. From this study, the goal is to establish that the investigational extended 2-dose regimens (0, 12 months; 0, 24 months; 0, 36 months; and 0, 60 months) studied in boys and girls 9 to 14 years of age are generally safe and immunogenic, with an antibody response that is not inferior to that observed in young women 16 to 26 years of age who receive the standard 3-dose regimen of 9-valent human papillomavirus (9vHPV) vaccine at 0, 2, and 6 months (i.e., the population and dose regimen used to establish 9vHPV vaccine efficacy).

ELIGIBILITY:
Inclusion Criteria:

Boys and Girls 9 to 15 Years:

- Must not have had coitarche and does not plan on becoming sexually active during the vaccination period

Women 16 to 26 Years:

* Has never had a Papanicolaou (Pap) test or only had normal Pap test results
* A lifetime history of 0 to 4 male and/or female sexual partners

Cohort 0 Participants:

- Received 1 dose of 9vHPV vaccine at least 1 year prior to enrollment and did not receive a second dose of any HPV vaccine

Exclusion Criteria:

All Participants:

* Known allergy to any vaccine component
* History of severe allergic reaction that required medical intervention
* Thrombocytopenia or any coagulation disorder
* Females only: participant is pregnant or expecting to donate eggs during day 1 through month 7
* Currently immunocompromised, or been diagnosed with immunodeficiency
* Had a splenectomy
* Receiving or has received immunosuppressive therapies within the last year
* Received any immunoglobulin product or blood-derived product within 3 months
* Has received more than 1 dose of an HPV vaccine (Cohort 0)
* Received a marketed HPV vaccine or has participated in an HPV vaccine clinical trial (Cohorts 1-5)

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Healthy male and female participants between the ages of 9 to 15 years (inclusive) and female participants between the ages of 16 and 26 years (inclusive) will be enrolled in this study.
Enrollment: 700 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2029-10-23 (Estimated); Study Completion 2029-10-23 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titers of Anti-Human Papilloma Virus Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 as Measured by Competitive Luminex Immunoassay | 4 weeks post last vaccination (Up to ~Month 61)
  Serum antibody titers for human papilloma virus (HPV) types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using competitive luminex immunoassay (cLIA). The geometric mean titer (GMT) for each HPV type will be reported in milli Merck units/mL (mMU/mL).
Percentage of Participants With at Least 1 Solicited Injection-site Adverse Event | Up to 5 days post vaccination
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants with injection-site AEs (erythema/redness, pain and swelling) will be assessed.
Percentage of Participants With at Least 1 Systemic Adverse Event | Up to 15 days post vaccination
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants with a systemic AE will be assessed.
Percentage of Participants With at Least 1 Serious Vaccine-Related Adverse Event | Entire study period (Up to ~Month 96)
  A serious adverse event (SAE) is defined as one that results in death, is life threatening, or requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or other important medical event that may require medical intervention. An SAE that is judged by the investigator to be related to the study vaccine is defined as a vaccine-related SAE.

SECONDARY OUTCOMES:
Percentage of Participants (Cohorts 1 to 5) Who Are Seropositive for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 4 weeks post last vaccination
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The percentage of participants who are seropositive (analysis population Cohorts 1 through 5 only) for each HPV type will be assessed.
Geometric Mean Titers (Cohorts 1 to 5) of Anti HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 12 months post last vaccination
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type (analysis population Cohorts 1 through 5 only) will be reported in mMU/mL.
Percentage of Participants (Cohorts 1 to 5) Who Are Seropositive for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 12 months post last vaccination
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The percentage of participants who are seropositive (analysis population Cohorts 1 through 5 only) for each HPV type will be assessed.
Geometric Mean Titers ( Cohorts 1 to 5) of Anti HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 24 months post last vaccination
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type (analysis population Cohorts 1 through 5 only) will be reported in mMU/mL.
Percentage of Participants (Cohorts 1 to 5) Who Are Seropositive for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 24 months post last vaccination
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The percentage of participants who are seropositive (analysis population Cohorts 1 through 5 only) for each HPV type will be assessed.
Geometric Mean Titers ( Cohorts 1 to 5) of Anti HPV Types 6, 11, 16, 18, 31, 33, 45, 52 , and 58 | 36 months post last vaccination
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The GMT for each HPV type (analysis population Cohorts 1 through 5 only) will be reported in mMU/mL.
Percentage of Participants (Cohorts 1 to 5) Who Are Seropositive for HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | 36 months post last vaccination
  Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52 and 58 will be determined using cLIA. The percentage of participants who are seropositive (analysis population Cohorts 1 through 5 only) for each HPV type will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (30):
- United States (14):
  - Kaiser Permanente Daly City ( Site 0044), Daly City, California
  - Kaiser Permanente Oakland ( Site 0020), Oakland, California
  - Kaiser Permanente Roseville ( Site 0047), Roseville, California
  - Kaiser Permanente Sacramento ( Site 0043), Sacramento, California
  - Kaiser Permanente South Sacramento ( Site 0045), Sacramento, California
  - Kaiser Permanente San Jose ( Site 0046), San Jose, California
  - Kaiser Permanente Santa Clara ( Site 0042), Santa Clara, California
  - Encompass Clinical Research ( Site 0022), Spring Valley, California
  - Advanced Research for Health Improvement, LLC-Pediatrics ( Site 0007), Naples, Florida
  - Tribe Clinical Research, LLC ( Site 0010), Greenville, South Carolina
  - Coastal Carolina Research Center ( Site 0032), North Charleston, South Carolina
  - Coastal Bend Clinical Research ( Site 0025), Corpus Christi, Texas
  - University of Texas Medical Branch-Sealy Institute for Vaccine Sciences Clinical Trials Program ( Si, Galveston, Texas
  - MultiCare Rockwood Cheney Clinic ( Site 0038), Cheney, Washington
- Colombia (2):
  - Fundación Centro de Investigación Clínica CIC ( Site 0157), Medellín, Antioquia
  - Centro de Atención e Investigación Médica SAS - CAIMED CHIA ( Site 0151), Chía, Cundinamarca
- Mexico (4):
  - CAIMED México ( Site 0207), Mexico City, Mexico City
  - AINPAD ( Site 0204), Morelia, Michoacán
  - Unidad biomedica avanzada monterrey ( Site 0203), Monterrey, Nuevo León
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan (, Mérida, Yucatán
- Poland (4):
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska ( Site 0557), Tarnów, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny-Klinika Pediatrii i Chorob Infekcyjnych ( Site 0556), Wroclaw, Lower Silesian Voivodeship
  - Jerzy Brzostek Prywatny Gabinet Lekarski ( Site 0553), Dębica, Podkarpackie Voivodeship
  - Gravita Diagnostyka i Leczenie Nieplodnosci ( Site 0555), Lodz, Łódź Voivodeship
- South Africa (3):
  - Perinatal HIV Research Unit_Do not use - Duplicate facility ( Site 0351), Johannesburg, Gauteng
  - TREAD Research ( Site 0354), Cape Town, Western Cape
  - Desmond Tutu HIV Foundation ( Site 0355), Cape Town, Western Cape
- Taiwan (3):
  - Taichung Veterans General Hospital ( Site 0653), Taichung
  - National Taiwan University Hospital ( Site 0651), Taipei
  - Chang Gung Medical Foundation.Linkou Branch ( Site 0652), Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Teppler H, Bautista O; Thomas Group; Flores S, McCauley J, Luxembourg A. Design of a Phase III immunogenicity and safety study evaluating two-dose regimens of 9-valent human papillomavirus (9vHPV) vaccine with extended dosing intervals. Contemp Clin Trials. 2021 Jun;105:106403. doi: 10.1016/j.cct.2021.106403. Epub 2021 Apr 12. PMID 33857679
- [Result] Klein NP, Wiesner A, Bautista O, Group T, Kanu K, Li ZL, McCauley J, Saxena K, Tota J, Luxembourg A, Bonawitz R. Immunogenicity and Safety of Extended-Interval 2-Dose Regimens of 9vHPV Vaccine. Pediatrics. 2024 Aug 1;154(2):e2023064693. doi: 10.1542/peds.2023-064693. PMID 38978512
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26176&tenant=MT_MSD_9011